CLINICAL TRIAL: NCT02375087
Title: Sleep Breathing Disorders, a Main Trigger for Cardiac ARythmias in Type I Myotonic Dystrophy ?
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: "STAR"
Record Dates: First submitted 2015-02-03; First posted 2015-03-02 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Up to one-third of patients with myotonic dystrophy type 1 die suddenly mainly from arrhythmias. Sleep apnea is prevalent in myotonic dystrophy (DM1) patients. Among the serious complications from sleep apnea, the most alarming are arrhythmias and sudden cardiac death (SCD). Diagnosis of sleep apnea using simple tools in ambulatory cardiology practice may improve therapy of cardiac arrhythmias in patients with DM1

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) and central sleep apnea (CSA), the most common form of sleep disordered breathing (SDB), are prevalent in patients with myotonic dystrophy type 1 (DM1). Among the serious complications from sleep apnea, the most alarming are cardiovascular, including arrhythmias and sudden cardiac death (SCD). Diagnosis of SDB using simple tools in ambulatory cardiology practice may lead to an important primary or additional therapy to supplement the use of drugs or devices in the treatment of cardiac arrhythmias.

We hypothesize that DM1 patients with severe oxygen desaturations (Oxygen desaturation index >15/hour of sleep and/or cumulative time spent below 90% of SaO2 above 5% of time of recording) will exhibit three fold more nocturnal arrhythmias compared to DM1 group without oxygen desaturations during sleep.

During this project we will address the following aims:

* Is there a relationship between the severity of oxygen desaturations during sleep and nocturnal arrhythmias? We will address this question in a prospective study with seven nights of at home recordings with a multimodal holter EKG assessing together arrhythmias, thoracic impedance (in order to estimate respiratory movements) and SaO2.
* The specific proarrhythmic role of REM sleep will be assessed during a single night full polysomnography and multiple sleep latency tests (MSLT).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from myotonic dystrophy (DM1)
* DM1 patients participating in the clinical cohorts of Grenoble, Saint-Etienne and Montpellier.
* Patients implanted or not with pacing devices or cardioverter-defibrillator (ICD).
* Patients treated or not by non invasive ventilation (NIV) at home. As a majority, of the patients with DM1 are poorly adherent with NIV they continue to exhibit significant desaturation during night. Truly compliant patients (mean daily duration>6/h night) will be studied as a predefined subgroup to assess the protective effect of NIV for suppressing oxygen desaturations and avoiding occurrence of nocturnal arrhythmias.

Exclusion Criteria:

* Patients who have had an acute episode of respiratory failure in the previous month
* Incapacitated patients in accordance with article L 1121-6 of the public health code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from myotonic dystrophy (DM1)
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Cardiac arythmia related to hypoxia and respiratory events | 7days
  Ambulatory at home concurrent assessment of arrhythmias and sleep breathing disorders by a multi-modal ECG Holter (Vista O2; Novacor, Rueil Malmaison, FranceTM). We will record seven consecutive nights at home to increase the sensitivity and the number of abnormal rhythmic events available for analysis. One night full polysomnography followed by Multiple sleep latency tests

SECONDARY OUTCOMES:
A temporal link between Sleep desordered breathing events and the developpement of arrythmias | 7 days
  More specifically the occurrence of arrhythmias will be correlated with the severity of oxygen desaturation
To assess during the entire night the increase in sympathetic activity (LF/HF ratio) in response to abnormal respiratory events during sleep and the relationship between sympathetic activity and prevalence of arrhythmias | 7 days
To compare arrhythmias prevalence in REM and non REM sleep | 7 days
To see whether a high adherence to non invasive ventilation (>6hours/night) and the suppression of oxygen desaturation is associated with a lower prevalence of arrhythmias | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Grenoble, France